CLINICAL TRIAL: NCT06675838
Title: The Effect of Time Management Training Based on Slavin's Effective Teaching Model on Procrastination Behavior in Nursing Students: a Quasi-Experimental Study
Brief Title: Impact of Slavin's Effective Teaching Model on Procrastination in Nursing Students: a Quasi-Experimental Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Seda Tugba Baykara Mat, Asst.Prof., University of Beykent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: The Effect of Time Management
Record Dates: First submitted 2024-10-31; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Procrastination; Educational Intervention; Time Management
Keywords: Procrastination; Academic Performance; Time Management; Nursing Students; Educational Intervention; Behavior Modification
MeSH Terms: interventions — Time Management

STUDY DESIGN:
Intervention Model Description: Intervention Content
  Training Program Name: Time Management and Procrastination Behavior Management Training Duration: 3 sessions of 1 hour each, 5-day program Target Audience: Intern Nurses
  Training Content:
  Fundamentals of Time Management:
  Definition and importance of time management. Fundamental principles for effective time use (prioritization, time blocking, planning).
  Understanding Procrastination Behavior:
  Definition and reasons for procrastination behavior. Effects of procrastination on student success.
  Time Management Strategies:
  Task Prioritization: Differentiating between urgent and important tasks. Time Blocking: Completing specific tasks in designated time slots. Daily Planning: Organizing daily tasks and activities.
  Managing Procrastination Behavior:
  Identification and analysis of procrastination habits. Coping strategies for procrastination (e.g., goal setting, increasing motivation, self-rewarding).
  Effective Teaching Techniques:
  Presentations and Information Sh
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nursing students (Experimental): Pre-Test and Post-Test Single Group Study
  Interventions: Behavioral: Time Management and Procrastination Behavior Management Training

INTERVENTIONS:
Behavioral: Time Management and Procrastination Behavior Management Training — Intervention Content
  Training Program Name: Time Management and Procrastination Behavior Management Training Duration: 3 sessions of 1 hour each, 5-day program Target Audience: Intern Nurses
  Training Content:
  Fundamentals of Time Management:
  Definition and importance of time management. Key principles for effective use of time (prioritization, time blocking, planning).
  Understanding Procrastination Behavior:
  Definition and reasons for procrastination behavior. Effects of procrastination on student success.
  Time Management Strategies:
  Task Prioritization: Differentiating between urgent and important tasks. Time Blocking: Completing specific tasks in designated time slots. Daily Planning: Organizing daily tasks and activities.
  Managing Procrastination Behavior:
  Identification and analysis of procrastination habits. Coping strategies for procrastination (e.g., goal setting, increasing motivation, self-rewarding).
  Effective Teaching Techniques:
  Presentations and Information Sharing

SUMMARY:
The purpose of this clinical trial is to determine if a time management training program can effectively reduce procrastination behavior among intern nursing students. It will also explore the impact of this training on students' academic performance and well-being. The main questions it aims to answer are:

Does the training reduce procrastination behavior in nursing students? How does the training impact time management skills and academic outcomes? Researchers will implement a time management training program based on the Effective Teaching Model to analyze changes in procrastination behavior.

Participants will:

Attend a five-day training program, with daily sessions covering specific topics on time management and procrastination Complete a pre-test and post-test to measure changes in procrastination behavior Provide feedback on the training program and engage in practical workshops The study will be conducted at a private university in Istanbul over a four-month period from November 2024 to March 2025, targeting all intern nursing students (N=70). Data will be collected using a general procrastination scale and analyzed for significant changes in time management and procrastination behaviors using SPSS software.

DETAILED DESCRIPTION:
Time management is a critical skill that directly affects success and efficiency in nursing students' educational processes. Procrastination can negatively impact both academic performance and the quality of clinical practice, making understanding and managing this behavior crucial for both students and healthcare services. This study aims to investigate the effects of a time management training program on procrastination behavior among intern nursing students. The training content, developed based on the Effective Teaching Model, will assess how students' time management skills and procrastination tendencies change. The study will be conducted at a private university in Istanbul from November 2024 to March 2025, with the target population being all intern nursing students enrolled at the university during the research period (N=70). No sampling will be done, and the aim is to reach the entire population.

The research aims to provide effective time management training for nursing students and to reduce procrastination behavior through this training. The training program will last for five days, with each day focusing on a specific topic. On the first day, the fundamentals of time management and understanding procrastination behavior will be covered. The second day will address time management strategies and techniques. The third day will focus on managing procrastination behavior and related strategies. On the fourth day, practical workshops will be conducted to create personal time management plans. The fifth day will include training evaluation, student feedback, and motivational activities. The training will utilize Slavin's Effective Teaching Model and will be enriched with presentations, interactive sessions, practical workshops, feedback, and motivational techniques. The program aims to enhance students' time management skills, reduce procrastination behavior, and improve academic performance. By the end of the training, a reduction in stress and anxiety levels, increased motivation, and overall improvement in quality of life are expected.

Data for the study will be collected using a personal information form and a general procrastination scale. Data analysis will be conducted using SPSS (Statistical Package for Social Sciences) for Windows 22.0. To determine if the research data follow a normal distribution, the Kolmogorov-Smirnov Test will be used. If p>0.05, the distribution is considered normal. If p<0.05, the distribution is not normal, and skewness and kurtosis values will be examined. Changes in repeated measurements will be analyzed using the repeated measures ANOVA test if the data are normally distributed, and the Friedman test if the data are not normally distributed. Initially, descriptive statistics will summarize the general characteristics of the data, and means and distributions of pre-test and post-test scores will be determined. The paired samples t-test will be used to evaluate differences between pre-test and post-test scores within the same group. This analysis will assess the impact of the training program on time management and procrastination behaviors. Additionally, effect size (e.g., Cohen's d) will be calculated to evaluate the magnitude and significance of the training intervention. Variance analysis (ANOVA) may be used to determine if there are significant differences between different groups, but its necessity will be determined based on the specifics of the study. Finally, power analysis will be performed to ensure the study's sample size is adequate. These analyses will collectively allow for meaningful and reliable interpretation of the research findings.

ELIGIBILITY:
Inclusion Criteria:

* Must be over 18 years of age.
* Must be registered as an intern nursing student at the university where the research is conducted.
* Must be attending full-time education.
* Must have a sufficient level of proficiency in understanding and speaking Turkish.
* Must be willing to participate voluntarily.

Exclusion Criteria:

* Change of department/school.
* Requesting to withdraw from the study.

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in Time Management Skills | Pre-test conducted one week prior to the training and post-test conducted immediately after the final training session.
  This outcome measure will evaluate the effectiveness of the "Time Management and Procrastination Behavior Management Training" on participants' time management skills. Participants will complete a standardized questionnaire assessing their self-reported time management abilities before and after the training to identify any significant changes.
  Student Information Form: This form consists of 8 questions regarding the socio-demographic information of immigrant students, including their country of origin, health status, and the healthcare institutions they have accessed.
  General Procrastination Scale: The General Procrastination Scale, developed by Çakıcı (2003), measures students' tendencies to procrastinate. The scale consists of 18 items rated on a 5-point Likert-type scale, and includes two subscales: "Procrastination" (items 2, 5, 7, 9, 10, 11, 13, 14, 15, 16, 18) and "Time Management" (items 1, 3, 4, 6, 8, 12, 17). Cronbach's alpha reliability coefficient was determined to be 0.81

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Beykent University, Istanbul, Beylikduzu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share Individual Participant Data (IPD) with other researchers. This decision is made to ensure the confidentiality and privacy of participants, as well as to maintain the integrity of the data collected for this specific study.